CLINICAL TRIAL: NCT03229213
Title: Evaluation of Physiological Responses During the Use of Interactive Video Game and the Cardiopulmonary Exercise Test in Cystic Fibrosis and Healthy Individuals
Brief Title: Interactive Video Game Responses in Cystic Fibrosis
Acronym: Igamecf
Status: Completed | Type: Observational
Sponsor: Pontificia Universidade Católica do Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Marcio Vinicius Fagundes Donadio, Professor, Pontificia Universidade Católica do Rio Grande do Sul
Other Study IDs: game
Record Dates: First submitted 2017-07-21; First posted 2017-07-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; video games; exercise; maximal oxygen consumption
MeSH Terms: conditions — Cystic Fibrosis; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cystic Fibrosis: Cystic fibrosis patients will be invited to participate in the study. All participants will complete a questionnaire to assess the level of physical activity prior to evaluation. On the first visit they will perform the cardiopulmonary exercise test (CPET) to evaluate cardiorespiratory responses during exercise. On the second visit an evaluation of the cardiorespiratory responses during the use of interactive video games (Nintendo Wii or Xbox One) will be performed. During interactive games, participants will use an accelerometer to assess the level of physical activity.
- Healthy: Healthy subjects will be invited to participate in the study. All participants will complete a questionnaire to assess the level of physical activity prior to evaluation. On the first visit they will perform the cardiopulmonary exercise test (CPET) to evaluate cardiorespiratory responses during exercise. On the second visit an evaluation of the cardiorespiratory responses during the use of interactive video games (Nintendo Wii or Xbox One) will be performed. During interactive games, participants will use an accelerometer to assess the level of physical activity.

SUMMARY:
Cystic fibrosis (CF) is a disease that affects multiple systems, however, the accumulation of secretion in the airways contributes to the fact that pulmonary complications are the main responsible for the high rates of morbidity and mortality. Physical exercise can be an important component in the treatment of these patients, and modalities such as Nintendo Wii and Xbox One stand out as feasible and innovative methods that can contribute to increase adherence to rehabilitation. Thus, the objective of this study is to compare the cardiorespiratory responses during a maximal exercise test with the use of Nintendo Wii and Xbox One in patients with CF and healthy individuals. Patients with a clinical diagnosis of CF, aged from 6 to 30 years old and in stable clinical conditions will be included. For healthy individuals, those who are considered healthy from the application of a health questionnaire and also aged from 6 to 30 years old will be included. Patients in both groups with cardiopathies, musculoskeletal diseases, neurological diseases or signs of pulmonary exacerbation will be excluded. Participants will complete a questionnaire to assess their level of physical activity. Afterwards, cardiopulmonary exercise test (CPET) will be performed (visit 1), followed by the use of video games (visit 2). The video game will be practiced using a Nintendo Wii and a Xbox One (10 minutes each). A rest of 10 minutes will be provided between the use of each video game. During the interactive games, patients will use an accelerometer to assess the level of physical activity. In parallel to this, healthy subjects will be invited to perform the same tests in two visits. To evaluate the perception of fatigue, the OMNI scale will be used. In addition, individuals will be asked to evaluate their level of satisfaction after each game.

DETAILED DESCRIPTION:
Cardiopulmonary exercise test: The test will be performed according to the recommendations of the American Thoracic Society and American College of Chest Physician.The variables to be measured includes maximal oxygen uptake (VO2max), maximal ventilation (Vemax), respiratory quotient (RQ), peripheral oxygen saturation (SpO2), subjective levels of dyspnea and fatigue in the legs (modified BORG scale), pulse oxygen (VO2/HR) and maximal heart rate (HRmax). During the test, the individuals will be asked to walk for 2 minutes to adapt to the treadmill, with a speed of 3 km/h and without inclination. After that, there will be increments in the speed of 0.5 Km/h, every minute, with a fixed slope of 3%, until the end of the test. All individuals will be encouraged to keep the pace until signs of exhaustion or limiting symptoms appear (dyspnea, leg pain and/or dizziness). To be considered a maximal test, at least three of the following criteria should be observed: exhaustion or inability to maintain the required speed, RQ>1.10, maximal achieved HR>85% of the estimated HR (formula: 220- Age) and the presence of a plateau in the VO2max.

Interactive Video Games: Participants will use Nintendo Wii for 10 minutes and then use Xbox One for 10 minutes, taking a 10-minute rest between one console and another. During the two video games, patients will use a Neoprene mask to collect gases, including maximal oxygen (VO2), carbon dioxide (CO2), maximal ventilation (VEmax), respiratory quotient (RQ) and the metabolic equivalents for oxygen (VE/VO2) and for carbon dioxide (VE/VCO2). In addition, peripheral oxygen saturation (SpO2), subjective levels of dyspnea and fatigue in the legs (modified BORG scale), pulse oxygen (VO2/HR) and maximal heart rate (HRmax) before and after Intervention will be collected.

Accelerometer: All participants will use an accelerometer while playing in the interactive video games. This equipment will be used on the left side of the waist. The results of the physical activity variables will be expressed as mean counts/min, as a mean indicator of the intensity of physical activity. In addition, the time spent in activities according to their intensity will be classified as sedentary (<100 counts), mild (≥100 counts) and moderate to vigorous (>2296 counts).

Scales: In the OMNI scale, individuals point out on a scale of 0 to 10 the fatigue level, where 0 is very easy and 10 is very difficult.Also, the level of satisfaction will be evaluated using a 5-point Likert scale where 1 represents no satisfaction and 5 much satisfaction.

ELIGIBILITY:
Inclusion Criteria:

Cystic fibrosis - clinical diagnosis of cystic fibrosis confirmed by sweat test or genetic test, aged from 6 to 30 years old and presenting stable clinical conditions.

Healthy individuals - to be considered healthy from the application of the health questionnaire and aged from 6 to 30 years old.

Exclusion Criteria:

Patients in both groups who present with cardiopathies, musculoskeletal diseases, neurological diseases or signs of pulmonary exacerbation will be excluded from the study. In addition, those subjects who have difficulty in understanding or are unable to perform the cardiopulmonary exercise test will also be excluded.

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients with cystic fibrosis, recruited at the CF center of Hospital São Lucas (PUCRS), and healthy individuals recruited from the loccal community.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Maximal oxygen consumption | Immediately after test or game
  Maximal oxygen consumption will be assessed during a maximal cardiopulmonary exercise test and during de use of interactive video games.
Maximal heart rate | Immediately after test or game
  Maximal heart rate will be measured using a heart monitor

SECONDARY OUTCOMES:
Satisfaction | Immediately after games
  Satisfaction will be evaluated using a 5 point likert scale where 1 represents no satisfaction and 5 much satisfaction.
Physical activity levels | Immediately after games
  Physical activity levels will be evaluated using the accelerometer on the left side of the waist.
Subjective evaluation of dyspnea | Immediately after test or game
  Dyspnea will be evaluated using the modified BORG scale where 0 is no dyspnea and 10 is maximal dyspnea.
Perception of fatigue | Immediately after games
  Perception of fatigue will be evaluated using the OMNI scale where 0 is very easy and 10 is very difficult.
The peripheral oxygen saturation (SpO2) | Immediately after test or game
  The peripheral oxygen saturation will be evaluated using a pulse oximetry.
Maximal ventilation (VEmax) | Immediately after test or game
  Maximal ventilation (VEmax) will be evaluated using a computerized system coupled to a gas analyzer.
Respiratory quotient (RQ) | Immediately after test or game
  The respiratory quotient (RQ) will be evaluated using a computerized system coupled to a gas analyzer.
Metabolic equivalents for oxygen (VE/VO2) | Immediately after test or game
  Metabolic equivalents for oxygen will be evaluated using a computerized system coupled to a gas analyzer.
Metabolic equivalents for carbon dioxide (VE/VCO2) | Immediately after test or game
  Metabolic equivalents for carbon dioxide Metabolic equivalents for oxygen will be evaluated using a computerized system coupled to a gas analyzer.

CONTACTS AND LOCATIONS:
Overall Officials: Marcio Donadio, PhD, Principal Investigator — Pontificia Universidade Católica do Rio Grande do Sul
Locations (1):
- Pontifífia Universidade Católica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bradley JM, Moran FM, Elborn JS. Evidence for physical therapies (airway clearance and physical training) in cystic fibrosis: an overview of five Cochrane systematic reviews. Respir Med. 2006 Feb;100(2):191-201. doi: 10.1016/j.rmed.2005.11.028. PMID 16412951
- [Result] Main E. What is the best airway clearance technique in cystic fibrosis? Paediatr Respir Rev. 2013 May;14 Suppl 1:10-2. doi: 10.1016/j.prrv.2013.01.008. Epub 2013 Mar 26. PMID 23541002
- [Result] Robinson M, Bye PT. Mucociliary clearance in cystic fibrosis. Pediatr Pulmonol. 2002 Apr;33(4):293-306. doi: 10.1002/ppul.10079. PMID 11921459
- [Result] Hamosh A, FitzSimmons SC, Macek M Jr, Knowles MR, Rosenstein BJ, Cutting GR. Comparison of the clinical manifestations of cystic fibrosis in black and white patients. J Pediatr. 1998 Feb;132(2):255-9. doi: 10.1016/s0022-3476(98)70441-x. PMID 9506637
- [Result] Grasemann H, Stehling F, Brunar H, Widmann R, Laliberte TW, Molina L, Doring G, Ratjen F. Inhalation of Moli1901 in patients with cystic fibrosis. Chest. 2007 May;131(5):1461-6. doi: 10.1378/chest.06-2085. PMID 17494794
- [Result] Boucher RC. Evidence for airway surface dehydration as the initiating event in CF airway disease. J Intern Med. 2007 Jan;261(1):5-16. doi: 10.1111/j.1365-2796.2006.01744.x. PMID 17222164
- [Result] Rosenstein BJ, Langbaum TS. Incidence of distal intestinal obstruction syndrome in cystic fibrosis. J Pediatr Gastroenterol Nutr. 1983 May;2(2):299-301. PMID 6553601
- [Result] Salonini E, Gambazza S, Meneghelli I, Tridello G, Sanguanini M, Cazzarolli C, Zanini A, Assael BM. Active Video Game Playing in Children and Adolescents With Cystic Fibrosis: Exercise or Just Fun? Respir Care. 2015 Aug;60(8):1172-9. doi: 10.4187/respcare.03576. Epub 2015 Apr 21. PMID 25899477
- [Result] Lester MK, Flume PA. Airway-clearance therapy guidelines and implementation. Respir Care. 2009 Jun;54(6):733-50; discussion 751-3. doi: 10.4187/002013209790983205. PMID 19467161
- [Result] Marks JH. Airway clearance devices in cystic fibrosis. Paediatr Respir Rev. 2007 Mar;8(1):17-23. doi: 10.1016/j.prrv.2007.02.003. Epub 2007 Mar 21. PMID 17419974
- [Result] Smyth AR, Bell SC, Bojcin S, Bryon M, Duff A, Flume P, Kashirskaya N, Munck A, Ratjen F, Schwarzenberg SJ, Sermet-Gaudelus I, Southern KW, Taccetti G, Ullrich G, Wolfe S; European Cystic Fibrosis Society. European Cystic Fibrosis Society Standards of Care: Best Practice guidelines. J Cyst Fibros. 2014 May;13 Suppl 1:S23-42. doi: 10.1016/j.jcf.2014.03.010. PMID 24856775
- [Result] Pinet C, Scillia P, Cassart M, Lamotte M, Knoop C, Melot C, Estenne M. Preferential reduction of quadriceps over respiratory muscle strength and bulk after lung transplantation for cystic fibrosis. Thorax. 2004 Sep;59(9):783-9. doi: 10.1136/thx.2004.021766. PMID 15333856
- [Result] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Result] O'Donovan C, Greally P, Canny G, McNally P, Hussey J. Active video games as an exercise tool for children with cystic fibrosis. J Cyst Fibros. 2014 May;13(3):341-6. doi: 10.1016/j.jcf.2013.10.008. Epub 2013 Nov 1. PMID 24189057
- [Result] American College of Sports Medicine Position Stand. The recommended quantity and quality of exercise for developing and maintaining cardiorespiratory and muscular fitness, and flexibility in healthy adults. Med Sci Sports Exerc. 1998 Jun;30(6):975-91. doi: 10.1097/00005768-199806000-00032. PMID 9624661
- [Result] Rand S, Hill L, Prasad SA. Physiotherapy in cystic fibrosis: optimising techniques to improve outcomes. Paediatr Respir Rev. 2013 Dec;14(4):263-9. doi: 10.1016/j.prrv.2012.08.006. Epub 2012 Nov 4. PMID 24209461
- [Result] Kuys SS, Hall K, Peasey M, Wood M, Cobb R, Bell SC. Gaming console exercise and cycle or treadmill exercise provide similar cardiovascular demand in adults with cystic fibrosis: a randomised cross-over trial. J Physiother. 2011;57(1):35-40. doi: 10.1016/S1836-9553(11)70005-4. PMID 21402328
- [Result] del Corral T, Percegona J, Seborga M, Rabinovich RA, Vilaro J. Physiological response during activity programs using Wii-based video games in patients with cystic fibrosis (CF). J Cyst Fibros. 2014 Dec;13(6):706-11. doi: 10.1016/j.jcf.2014.05.004. Epub 2014 Jun 13. PMID 24935613
- [Result] Thompson PD, Arena R, Riebe D, Pescatello LS; American College of Sports Medicine. ACSM's new preparticipation health screening recommendations from ACSM's guidelines for exercise testing and prescription, ninth edition. Curr Sports Med Rep. 2013 Jul-Aug;12(4):215-7. doi: 10.1249/JSR.0b013e31829a68cf. No abstract available. PMID 23851406
- [Result] Rodrigues AN, Perez AJ, Carletti L, Bissoli NS, Abreu GR. Maximum oxygen uptake in adolescents as measured by cardiopulmonary exercise testing: a classification proposal. J Pediatr (Rio J). 2006 Nov-Dec;82(6):426-30. doi: 10.2223/JPED.1533. Epub 2006 Sep 21. PMID 17003945
- [Result] Karila C, de Blic J, Waernessyckle S, Benoist MR, Scheinmann P. Cardiopulmonary exercise testing in children: an individualized protocol for workload increase. Chest. 2001 Jul;120(1):81-7. doi: 10.1378/chest.120.1.81. PMID 11451820
- [Result] Higgins LW, Robertson RJ, Kelsey SF, Olson MB, Hoffman LA, Rebovich PJ, Haile L, Orenstein DM. Exercise intensity self-regulation using the OMNI scale in children with cystic fibrosis. Pediatr Pulmonol. 2013 May;48(5):497-505. doi: 10.1002/ppul.22639. Epub 2012 Sep 19. PMID 22997144
- [Result] Hallal PC, Reichert FF, Clark VL, Cordeira KL, Menezes AM, Eaton S, Ekelund U, Wells JC. Energy expenditure compared to physical activity measured by accelerometry and self-report in adolescents: a validation study. PLoS One. 2013 Nov 4;8(11):e77036. doi: 10.1371/journal.pone.0077036. eCollection 2013. PMID 24223707
- [Result] Evenson KR, Catellier DJ, Gill K, Ondrak KS, McMurray RG. Calibration of two objective measures of physical activity for children. J Sports Sci. 2008 Dec;26(14):1557-65. doi: 10.1080/02640410802334196. PMID 18949660